CLINICAL TRIAL: NCT01598506
Title: Determination of the ED50 of Intrathecal Hydromorphone in Laboring Women Using the Up-and-down Sequential Allocation Method
Brief Title: Intrathecal Hydromorphone for Labor Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Grant Lynde, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054701
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydromorphone (Experimental): Laboring patients receive ED50 of hydromorphone one time intrathecally
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone will be administered one time intrathecally to laboring patients to determine the ED50 for pain relief.

SUMMARY:
This study will investigate the dose of hydromorphone which will relieve the pain of women in labor when delivered directly in the area around the spinal cord (i.e., intrathecal injection). The primary objective is to determine the dose of intrathecal hydromorphone that results in a pain score of less than 4 out of 10 thirty minutes after intrathecal injection in 50% of women. Secondary objectives include determining this dose at five and ten minutes after injection. Thirty women admitted to labor and delivery for planned vaginal delivery desiring epidural placement will be consented for the study. The starting dose of intrathecal hydromorphone will be 6 mcg. The up-and-down sequential allocation method of statistical analysis will be used, meaning that each subsequent dose will be dependent upon the result obtained from the prior dose - ergo, if the initial subject has pain relief, the second subject will receive 4 mcg (2 mcg less), but if the initial subject does not have pain relief, the second subject will receive 8 mcg (2 mcg more) of hydromorphone.

After the intrathecal injection is given and the epidural is placed, visual analogue pain scores will be assessed 60 minutes following injection. A pain score of less than three will be a positive result. A pain score of three or greater will be a negative result. Blood pressure, heart rate, arterial oxygen saturation, fetal heart rate, and any side effects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Labor
* Desires pain relief

Exclusion Criteria:

* Any comorbidities other than obesity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant C Lynde, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] O'Reilly-Shah V, Lynde GC. Determination of ED50 and time to effectiveness for intrathecal hydromorphone in laboring patients using Dixon's up-and-down sequential allocation method. BMC Anesthesiol. 2018 Oct 5;18(1):140. doi: 10.1186/s12871-018-0603-8. PMID 30290794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled from January 2013 to November 2013
Groups:
- Hydromorphone: Laboring patients receive ED50 of hydromorphone one time intrathecally.
  ED50 of hydromorphone was 12.7 mcg +/- 3.27.
Period: Overall Study
Arm/Group | Hydromorphone
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hydromorphone
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain Score, Visual Analogue Pain Scores
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: 30 minutes after intrathecal injection
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Hydromorphone: Laboring patients receive ED50 of hydromorphone one time intrathecally.
  ED50 of hydromorphone was 10.9 (95% CI +/- 1.2 mcg).
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 1.9 [0 to 4]

2. Secondary Outcome: Pain Scores, Visual Analogue Pain Scale
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain).
Time Frame: Baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 20
units on a scale | 8.6 [7 to 10]

ADVERSE EVENTS:
Arm/Group | Hydromorphone
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes